CLINICAL TRIAL: NCT01304147
Title: Intranasal (IN) Ketamine in Treatment-Resistant Depression (TRD)
Brief Title: Intranasal Ketamine in Treatment-Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 11-0492; INKET-001
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Major Depressive Disorder
Keywords: ketamine; depression; treatment resistance; intranasal, antidepressant; glutamate; NMDA receptor
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Subjects randomized to this arm will receive the active study medication, intranasal ketamine.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive intranasal saline.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ketamine — A single dose of intranasal ketamine up to 50 mg
  Arms: Ketamine
Drug: placebo — Single dose of saline intranasal
  Arms: Placebo

SUMMARY:
The objective of the current study is to investigate the safety and efficacy of a single dose of intranasal (IN) ketamine in treatment-resistant depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21-65 years;
2. Women of childbearing potential must agree to use a medically accepted means of contraception for the duration of the study;
3. Primary diagnosis of major depressive disorder as assessed by the SCID-P;
4. Current depressive episode;
5. History of a failure to respond to at least one (1) adequate pharmacotherapy trials in the current major depressive episode;
6. Subjects must have scored ≥ 30 on the IDS-C30 at Screening ≥ 24 at Treatment Day #1 and #2;
7. Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document;
8. Subjects must be able to identify a family member, physician, or friend who will participate in the Treatment Contract and serve as an emergency contact.

Exclusion Criteria:

1. Women who plan to become pregnant, are pregnant or are breast-feeding;
2. Any unstable medical illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease;
3. Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
4. Lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, OCD, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
5. Drug or alcohol abuse or dependence within the preceding 6 months;
6. Lifetime abuse or dependence on ketamine or phencyclidine;
7. Patients judged by study investigator to be at high risk for suicide.
8. Previous participation in a ketamine study at Mount Sinai

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Lapidus KA, Levitch CF, Perez AM, Brallier JW, Parides MK, Soleimani L, Feder A, Iosifescu DV, Charney DS, Murrough JW. A randomized controlled trial of intranasal ketamine in major depressive disorder. Biol Psychiatry. 2014 Dec 15;76(12):970-6. doi: 10.1016/j.biopsych.2014.03.026. Epub 2014 Apr 3. PMID 24821196
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from physician referrals, media advertisements, and an academic outpatient psychiatric clinic. All study treatments were performed at Mount Sinai Medical Center between April 2012 and June 2013.
Groups:
- Ketamine Then Placebo: Ketamine: A single dose of intranasal ketamine up to 50 mg for 7 days in first intervention. Then Placebo for 7 days in 2nd intervention.
- Placebo, Then Ketamine: placebo: Single dose of saline (0.9% saline solution) intranasal for 7 days in first intervention, then Ketamine 50mg in second intervention.
Period: First Intervention (7days)
Arm/Group | Ketamine Then Placebo | Placebo, Then Ketamine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (1 Day)
Arm/Group | Ketamine Then Placebo | Placebo, Then Ketamine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (7days)
Arm/Group | Ketamine Then Placebo | Placebo, Then Ketamine
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: one participant data information missing for history of Psychotherapy, and history of Failed Antidepressant Medications.
Arm/Group | Participants Treated
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment
  years | 48.0 (12.8)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Married [Number; unit: participants]
  yes | 6
  no | 14
Employed [Number; unit: participants]
  yes | 10
  no | 10
Age of Onset [Mean (Standard Deviation); unit: years] | 21.4 (12.0)
Illness Duration in Years [Mean (Standard Deviation); unit: years] | 27.4 (13.7)
Chronic [Number; unit: participants]
  yes | 9
  no | 11
Recurrent [Number; unit: participants]
  yes | 17
  no | 3
Length of Current Episode in Years [Mean (Standard Deviation); unit: years] | 15.2 (17.4)
Failed Antidepressants Medications [Mean (Standard Deviation); unit: number of medications] — n=19 missing information for one participant
  number of medications | 4.1 (3.9)
History of Electroconvulsive Therapy [Number; unit: participants]
  yes | 4
  no | 16
History of Psychotherapy [Number; unit: participants] — n=19 missing information for one participant
  participants
    yes | 17
    no | 2
    missing information | 1
History of Suicide Attempts [Number; unit: participants]
  yes | 2
  no | 18
Past Substance Use Disorder [Number; unit: participants]
  yes | 3
  no | 17
Current Anxiety Disorder [Number; unit: participants]
  yes | 4
  no | 16
Melancholic [Number; unit: participants]
  yes | 9
  no | 11
Atypical [Number; unit: participants]
  yes | 2
  no | 18
Baseline Inventory of Depressive Symptoms- Clinician Rated (Screen) [Mean (Standard Deviation); unit: units on a scale] — Inventory of Depressive Symptoms - Clinician Rated (IDS-C) has 30 items. Each item is rated 0-3, total score rage from 0 to 90, from mild to severe.
  units on a scale | 42.7 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Number of patients meeting response criteria of >=50% decrease in MADRS score from baseline , ie, difference in depressive symptoms using MADRS instrument, 24 hours following drug administration
  10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 and 60 points.
Time Frame: 24 hours
Population: 20 patients randomized and 18 completed both treatment periods
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 18 | 18
participants | 8 | 1
Statistical Analysis 1: Comparison: Ketamine vs Placebo; within-subject crossover design; Test type: Superiority or Other; p < 0.001, Paired t-test, 2 sided; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [3.9 to 11.3]

2. Secondary Outcome: Systematic Assessment for Treatment Emergent Effects (SAFTEE)
Description: This is a self-report measure for systematically assessing 48 possible adverse events. It documents their severity, relationship to study drug, and the action taken.
Time Frame: 2 weeks
Population: Number of events, more detailed in adverse event section
Measure: Number; unit: events
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 19 | 19
events | 79 | 57

ADVERSE EVENTS:
Time Frame: within 24 hours following treatment
Description: No serious adverse events occurred during the study.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=19) | Placebo (N=19)
Feeling strange or unreal (General disorders) | 8 (8) | 0 (0)
Poor Memory (General disorders) | 7 (7) | 2 (2)
Weakness or fatigue (General disorders) | 6 (6) | 1 (1)
Delayed or absent orgasm (Social circumstances) | 5 (5) | 0 (0)
Loss of sexual interest (Social circumstances) | 4 (4) | 1 (1)
Trouble concentrating (General disorders) | 4 (4) | 2 (2)
Problems with sexual arousal (Social circumstances) | 4 (4) | 3 (3)
Dizziness or fainting (General disorders) | 3 (3) | 0 (0)
Dizziness when you stand up (General disorders) | 3 (3) | 2 (2)
Diminished mental (Psychiatric disorders) | 3 (3) | 3 (3)
Feeling drowsy or sleepy (General disorders) | 3 (3) | 4 (4)
Poor coordination or unsteadiness (General disorders) | 3 (3) | 0 (0)
Difficulties finding words (General disorders) | 3 (3) | 2 (2)
Abnormal sensations (General disorders) | 2 (2) | 0 (0)
Numbness or tingling (General disorders) | 2 (2) | 0 (0)
Strange taste in mouth (General disorders) | 2 (2) | 1 (1)
Nightmares or other sleep disturbance (General disorders) | 2 (2) | 5 (5)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Appetite decreased (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Heartbeat rapid or pounding (General disorders) | 1 (1) | 1 (1)
Clenching of teeth at night (General disorders) | 1 (1) | 1 (1)
Stuffy nose (General disorders) | 1 (1) | 2 (2)
Irritable (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Tremor or shakiness (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Trouble sitting still (General disorders) | 1 (1) | 1 (1)
Feeling nervous or hyper (General disorders) | 1 (1) | 2 (2)
Frequent need to urinate (Renal and urinary disorders) | 1 (1) | 2 (2)
Apathy/Emotional indifference (General disorders) | 1 (1) | 2 (2)
Trouble sleeping (General disorders) | 1 (1) | 9 (9)
Muscle twitching or movements (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach or abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appetite increased (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ringing in ears or trouble hearing (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Unable to sit still (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size. Ongoing treatment with psychotropic medication allowed at stable doses makes it difficult to distinguish an intrinsic effect of ketamine from benefits resulting from the combination of ketamine with other antidepressant agents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes